CLINICAL TRIAL: NCT06523309
Title: Prospective Registry of Electroacupuncture Treatment for Patients With Different Behavioral and Psycological Symptoms of Alzheimer's Disease
Brief Title: Electroacupuncture Treatment of Behavioral and Psycological Symptoms in Patients With Alzheimer's Disease
Status: Not yet recruiting | Type: Observational
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Bao-Hui Jia, Director of rehabilitation Medicine, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Other Study IDs: 2024-076-KY-01
Record Dates: First submitted 2024-07-19; First posted 2024-07-26 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: BPSD (Behavioral and Psycological Symptoms of Dementia); Alzheimer's Dementia
MeSH Terms: conditions — Behavior; Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Affective symptom group: A group of Alzheimer's patients showing emotional symptoms such as anxiety, depression, apathy, etc.
  Interventions: Other: Electroacupuncture treatment
- Psychotic symptom group: A group of Alzheimer's patients showing psychotic symptoms such as delusions, hallucinations, etc.
  Interventions: Other: Electroacupuncture treatment
- Hyperactivity symptom group: A group of Alzheimer's patients showing hyperactivity symptoms such as irritability, aggression, aberrant motor behaviour, etc.
  Interventions: Other: Electroacupuncture treatment
- Euphoric symptom group: A group of Alzheimer's patients showing euphpric symptoms.
  Interventions: Other: Electroacupuncture treatment

INTERVENTIONS:
Other: Electroacupuncture treatment — Electroacupuncture treatment consists of conventional acupuncture and electrical stimulation. After acupuncture, the electrical stimulation is continuously stimulated.

SUMMARY:
This study aims to establish a prospective case registration research platform for electroacupuncture in treating behavioral and psychological symptoms in patients with mild to moderate Alzheimer's disease, and to investigate the dose-effect relationship and cost-effectiveness of electroacupuncture for these symptoms.

DETAILED DESCRIPTION:
To establish a prospective case registration research platform aimed at treating mild to moderate Alzheimer's disease patients presenting with behavioral and psychological symptoms. This platform will document the electroacupuncture treatment process, conduct regular assessments using neuropsychiatric questionnaires (NPI) and the Alzheimer's Disease Cooperative Study - Clinical Global Impression of Change Scale (ADAS-CGIC), and compare the effects of different parameters, treatment frequency, and duration of electroacupuncture on therapeutic outcomes for various behavioral and psychological symptoms in Alzheimer's disease patients. Furthermore, it aims to investigate the influencing factors of electroacupuncture treatment for behavioral and psychological symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the diagnostic criteria for AD in the NIA-AA standard;
2. Clinical dementia rating scale ≤2 points;
3. Accompanied by at least one psychobehavioral symptom, NPI：frequency × degree ≥1 point;
4. Sign informed consent.

Exclusion Criteria:

1.There are contraindications for acupuncture treatment, such as the tendency of acupoint bleeding or allergy to metal

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Alzheimer's disease patients with behavioral and psycological symptoms, such as apathy, depression, anxiety, delusions, hallucinations, irritability, etc.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-07-30 (Estimated); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Neuropsychiatric Inventory (NPI) | NPI will be performed before treatment and every month after treatment for up to 24 months
  NPI is used to evaluate neuropsychiatric behavioral symptoms of dementia patients. The scale assesses the neuropsychiatric disorders of patients according to the caregiver's view of the patient's behavior and the corresponding distress felt by the patient. The scoring range of the patient evaluation scale is 0-144 points, and the scoring of the caregiver distress scale is 0-60 points, the lower the score is, the better the patient's condition is.
Alzheimer's Disease Cooperative Study-Clinical Global Impression of Change (ADCS-CGIC) | The ADCS-CGIC will be performed before treatment and every 2 month after treatment for up to 24 months
  ADCS-CGIC is a global rating of change developed to assess clinically significant change in symptoms over time in AD clinical trials. Clinicians rate patient symptoms on the ADCS-CGIC as: very much improved (1), much improved (2), minimally improved (3), no change (4), minimally worse (5), much worse (6), and very much worse (7) compared to baseline symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Baohui Jia, Principal Investigator — Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Locations (7):
- China (7):
  - Beijing United Family Rehabilitation Hospital, Beijing, Beijing Municipality
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - Guang'anmen Hospital of China Academy of Chinese Medical Sciences, Beijing, Beijing Municipality
  - Xuanwu Hospital of Capital Medical University, Beijing, Beijing Municipality
  - Beijing Geriatric Hospital, Beijing, Beijing Municipality
  - Fujian University of Traditional Chinese Medicine, Fuzhou, Fujian
  - The Second Affiliated Hospital of Heilongjiang University of Chinese Medicine, Harbin, Heilongjiang

IPD SHARING:
Plan to Share IPD: No